CLINICAL TRIAL: NCT02001064
Title: Pilot Study of Care4Today v.2.0 Application for Improving Adherence to HIV Medications
Brief Title: Care4Today v2.0 Application for Improving Adherence to HIV Medications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Principal Investigator, David J. Moore, Ph.D., Professor of Psychiatry, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Care4Today-13
Record Dates: First submitted 2013-11-27; First posted 2013-12-04 (Estimated); Results first posted 2021-07-29 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: HIV; AIDS
Keywords: interventions; technology; adherence; ARV
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Care4Today v2.0 mobile application + electronic monitoring of adherence (Experimental): Care4Today v2.0 mobile application
  Participants in the experimental application arm will use the Care4Today v2.0 mobile application for antiretroviral medication adherence support. Alert messages generated via the app will be targeted to the specific schedule and needs of the individual.
  Electronic monitoring of adherence:
  Participants' adherence to antiretroviral therapy medication is measured via Medication Event Monitoring System (MEMS) cap.
  Interventions: Behavioral: Care4Today v2.0 mobile application + electronic monitoring of adherence
- Electronic monitoring of adherence (No Intervention): Participants' adherence to antiretroviral therapy medication is measured via Medication Event Monitoring System (MEMS) cap.

INTERVENTIONS:
Behavioral: Care4Today v2.0 mobile application + electronic monitoring of adherence — Care4Today mobile application will send automated medication alert messages to HIV-infected persons. The alert messages are customizable and automated, and real-time results are viewable within the application. The Care4Today intervention is designed to improve adherence to ART medications among HIV-infected persons who experience adherence difficulties over standard of care.
  Arms: Care4Today v2.0 mobile application + electronic monitoring of adherence

SUMMARY:
Although poor antiretroviral (ART) adherence in HIV does not mean a complete lack of therapeutic results, the benefit of ART increases as adherence improves. Consequences of suboptimal ART adherence are viral rebound, development of drug-resistant HIV strains, and more rapid progression to AIDS. Moreover, HIV-infected persons tend to have numerous co-occurring conditions and therefore take many medications making adherence to multiple drug regimens more difficult. A mobile application capable of improving medication adherence among HIV-infected persons would be highly useful.

The investigators propose an intervention study designed to address these potential mechanisms of nonadherence by utilizing the Care4Today v2.0 smartphone application (app). The current study is a small pilot Randomized Controlled Trial (RCT) comparing the smart phone application titled "Care4Today v2.0" versus standard of care to improve medication adherence to ART over a 4-week period with 60 HIV-infected participants.

The pilot RCT consists of 60 HIV-infected persons who are at risk for ART medication nonadherence. Using random assignment, 30 HIV-infected participants will be assigned to medication adherence improvement via "Care4Today" app as compared to 30 HIV-infected participants assigned standard of care.

The investigators will assess the effectiveness and acceptability of the app in improving objectively measured ART adherence (i.e., via medication event monitoring system caps) over a 4-week period via a pilot RCT with 30 HIV-infected persons assigned to the Care4Today intervention and 30 HIV-infected persons assigned to standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent
* 18 years or older at the time of enrollment
* HIV-infected
* Taking at least one medication to treat HIV illness
* Indication of medication nonadherence, or having a condition (e.g., active substance use, depression) that puts the individual at risk for medication non adherence
* Willingness to use electronic monitoring caps to track ART medication
* Willingness to respond to application alert messages

Exclusion Criteria:

* Axis I psychiatric diagnosis of psychotic disorder or mood disorder with psychotic features
* Presence of a neurological condition (beyond HIV infection) known to impact cognitive functioning (e.g., Huntington's Disease, Stroke)
* Unwillingness or inability to use electronic medication monitoring technology
* Unwillingness or inability to use daily alert messages

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J. Moore, Ph.D., Principal Investigator — University of California, San Diego
Locations (1):
- Hnrc-Tmarc, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: We enrolled 60 participants for the study cohort. 58 participants completed the initial assessment, 2 decided to discontinue after randomization (both did not wish to use the mobile application and phone for the duration of the study). Additionally, 1 participant decided to no longer participate in research studies between visits one and two.
Groups:
- Care4Today v2.0 Mobile Application + Electronic Monitoring of Adherence: Care4Today v2.0 mobile application
  Participants in the experimental application arm will use the Care4Today v2.0 mobile application for antiretroviral medication adherence support. Alert messages generated via the app will be targeted to the specific schedule and needs of the individual.
  Electronic monitoring of adherence:
  Participants' adherence to antiretroviral therapy medication is measured via MEMS cap.
- Electronic Monitoring of Adherence: Electronic monitoring of adherence:
  Participants' adherence to antiretroviral therapy medication is measured via MEMS cap.
Period: Overall Study
Arm/Group | Care4Today v2.0 Mobile Application + Electronic Monitoring of Adherence | Electronic Monitoring of Adherence
Started | 30 | 30
Completed | 28 | 29
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Care4Today v2.0 Mobile Application + Electronic Monitoring of Adherence | Electronic Monitoring of Adherence | Total
Number analyzed (Participants) | 28 | 29 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.8 (9.6) | 48.5 (9.5) | 49.2 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 24 | 27 | 51
Race/Ethnicity, Customized [Number; unit: participants]
  Non-Hispanic White | 14 | 15 | 29
  Non-Hispanic Black | 12 | 8 | 20
  Hispanic | 1 | 5 | 6
  Other | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 28 | 29 | 57
Education [Mean (Standard Deviation); unit: years] | 13.9 (2.2) | 12.9 (2.9) | 13.4 (2.6)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants ≥90% Adherent to Antiretroviral Medication Based on MEMS Cap Openings
Description: Adherence will be measured using Medication Event Monitoring Systems (MEMS). Adherence defined as % MEMS adherence (doses taken/doses prescribed) within 2 hours of the indicated dose time. Adherence was dichotomized into 2 groups: <90% and ≥90% using MEMS caps.
Time Frame: Completion of 30-day intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Care4Today v2.0 Mobile Application + Electronic Monitoring of Adherence | Electronic Monitoring of Adherence
Number analyzed (Participants) | 28 | 29
Participants | 9 | 5
Statistical Analysis 1: Comparison: Care4Today v2.0 Mobile Application + Electronic Monitoring of Adherence vs Electronic Monitoring of Adherence; Test type: Superiority; p = 0.32, t-test, 1 sided; Odds Ratio (OR) = 2.3

2. Primary Outcome: Average Minutes From Antiretroviral Medication Dose Time Based on MEMS Cap Openings
Description: The absolute value (in minutes) from the time a participant was scheduled to take an antiretroviral medication dose to when the participant opened the MEMS cap
Time Frame: Completion of 30-day intervention
Measure: Mean (Standard Deviation); unit: minutes from target dose time
Arm/Group | Care4Today v2.0 Mobile Application + Electronic Monitoring of Adherence | Electronic Monitoring of Adherence
Number analyzed (Participants) | 28 | 29
minutes from target dose time | 112.0 (112.0) | 146.7 (101.0)
Statistical Analysis 1: Comparison: Care4Today v2.0 Mobile Application + Electronic Monitoring of Adherence vs Electronic Monitoring of Adherence; Test type: Superiority; p = 0.073, Wilcoxon (Mann-Whitney) — Cohen's d (ranks) = -.049

3. Primary Outcome: Percentage of Doses Taken in Dose Time Window
Time Frame: Completion of 30-day intervention
Measure: Mean (Standard Deviation); unit: Percentage of doses taken in window
Arm/Group | Care4Today v2.0 Mobile Application + Electronic Monitoring of Adherence | Electronic Monitoring of Adherence
Number analyzed (Participants) | 28 | 29
Percentage of doses taken in window | 66.8 (27.0) | 57.5 (32.2)
Statistical Analysis 1: Comparison: Care4Today v2.0 Mobile Application + Electronic Monitoring of Adherence vs Electronic Monitoring of Adherence; Test type: Superiority; p = 0.24, Wilcoxon (Mann-Whitney) — Cohen's d=0.31

ADVERSE EVENTS:
Time Frame: Adverse event data were collected while participants were on study (i.e., 30 days)
Arm/Group | Care4Today v2.0 Mobile Application + Electronic Monitoring of Adherence | Electronic Monitoring of Adherence
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/29
Other Adverse Events (participants affected / at risk) | 0/28 | 0/28

LIMITATIONS AND CAVEATS:
1) Small sample size; 2) Short time period; 3) MEMS adherence data based on # of cap openings, not directly whether the medication was ingested; 4) No group without psychoeducation component

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No